CLINICAL TRIAL: NCT02299284
Title: Intensive Home-based Bimanual and Lower-limb Training in Young Children With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-219CR
Record Dates: First submitted 2014-11-12; First posted 2014-11-24 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cerebral Palsy
Keywords: Spastic; Hemiplegia
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hand-Arm Bimanual Intensive Therapy (HABIT) (Experimental): HABIT, bimanual training, bilateral training, restraint therapy, PT, OT, rehab
  Interventions: Other: Intensive Home-based Bimanual and Lower-limb Training in Young Children With Hemiplegia
- Intensive Functional Lower-Limb Training (Experimental): lower-limb function, strength training, balance, PT, OT, rehab
  Interventions: Other: Intensive Home-based Bimanual and Lower-limb Training in Young Children With Hemiplegia

INTERVENTIONS:
Other: Intensive Home-based Bimanual and Lower-limb Training in Young Children With Hemiplegia

SUMMARY:
A randomized control trial to test the efficacy of a new treatment involving intensive home-based bimanual training (Hand-Arm Bimanual Intensive Therapy (HABIT) and intensive home-based functional lower-limb training in children with hemiplegia. The protocols have been developed at TC Columbia University to be child friendly and draw upon the investigators experience since 1998 with intensive movement therapy in children with cerebral palsy. The aim is to promote either the use/coordination of movement of the hands or improve lower-limb balance, strength, and function. Caregivers will be trained at the investigator center and then be asked to do 2 hours per day, 5 days per week, for 9 weeks (90 hours total) of activities with their child in their own home. The activities will be supervised by the investigators team via computer. Participants do NOT need to live in the New York City area, but a one-time weekend visit to the investigators center is required for training. All measurement and treatment is performed in the home.

Participants are randomized to receive either HABIT or lower-limb training. If caregivers wish, they may chose to be crossed over at the end of the study and trained to receive the other treatment. PARTICIPATION IS FREE. Please check out the investigators website for more information: http://www.tc.edu/centers/cit/

DETAILED DESCRIPTION:
The investigators are currently recruiting children with hemiplegia between the ages of 2.5 to 12 years of age to participate in a study examining the effects of extensive practice on affected hand/arm use and lower- limb use. This is a research study that will teach caregivers how to administer either hand-arm bimanual intensive training (HABIT) or lower-limb intensive training in their own home. HABIT aims to improve the use and coordination of both arms in daily function, particularly during the performance of bimanual activities (i.e. buttoning a shirt, cutting with scissors). Lower-limb intensive training aims to improve the quality of lower-limb functioning with a particular focus on functional activities (i.e. getting up from a chair, walking, climbing stairs).

What does participation entail?

* Being randomized to learn to provide either intensive lower- or upper-limb activities in your own home (training will be provided over a a weekend session at our center)
* Getting trained to administer some basic upper- and lower-limb assessments in your own home
* Completing 90 hours of activities over a period of 9 weeks (2 hrs/day, 5 days/week; does not have to be 2 consecutive hours for daily activities)
* Videoconferencing online with a project supervisor at least 1 hour per week during activities
* Learning how to assess your child's motor function for posttesting.

Can I choose to receive upper or lower extremity training if my child qualifies?

• Unfortunately not, it must be randomly assigned as each group will be compared to the other. However, the investigators can provide training tips after completion of the study.

What if my child does not qualify?

* There may be opportunities at a later date or for another study.
* Please contact us at (212)-678-3332 or cpresearch@tc.columbia.edu if you have any questions.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 2.5 - 12 years with hemiplegia; hemiplegia due to result of prenatal stroke, brain lesion, or malformation (or within the two years of life).
* Children that have the ability to grasp or release objects with the affected hand
* Children who are able to walk independently without the assistance of a device
* Children that have the cognitive capability to follow simple instructions and interact in play activities 2 hours per day with a parent/caregiver.
* Caregivers willing to commit to the entire intervention period of 90 hours over 9 weeks
* Caregivers able to provide one-on-one attention to child during the daily two hours of activities (note: because this is part of a research study, we can only train one caregiver per household)

Exclusion Criteria:

* Children that have received Botox or are planning any new treatment within 6 mos. of enrollment in the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment | Change from baseline to 9 weeks
  measure of bimanual hand-use in spontaneous play setting
10 Meter walk test | Change from baseline to 9 weeks
  measures child's velocity when walking over 10 meters

SECONDARY OUTCOMES:
Assisting Hand Assessment | Change from baseline to 6 months
  measure of bimanual hand-use in spontaneous play setting
10 Meter walk test | Change from baseline to 6 months
  measures child's velocity when walking over 10 meters

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gordon, Ph.D., Study Director — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University Center for Cerebral Palsy Research, New York, New York, United States

REFERENCES:
- [Background] Charles J, Gordon AM. Development of hand-arm bimanual intensive training (HABIT) for improving bimanual coordination in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2006 Nov;48(11):931-6. doi: 10.1017/S0012162206002039. PMID 17044964
- [Result] Ferre CL, Brandao MB, Hung YC, Carmel JB, Gordon AM. Feasibility of caregiver-directed home-based hand-arm bimanual intensive training: a brief report. Dev Neurorehabil. 2015 Feb;18(1):69-74. doi: 10.3109/17518423.2014.948641. Epub 2014 Sep 2. PMID 25180530
- [Result] Gordon AM, Schneider JA, Chinnan A, Charles JR. Efficacy of a hand-arm bimanual intensive therapy (HABIT) in children with hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2007 Nov;49(11):830-8. doi: 10.1111/j.1469-8749.2007.00830.x. PMID 17979861
- [Derived] Surana BK, Ferre CL, Dew AP, Brandao M, Gordon AM, Moreau NG. Effectiveness of Lower-Extremity Functional Training (LIFT) in Young Children With Unilateral Spastic Cerebral Palsy: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2019 Oct;33(10):862-872. doi: 10.1177/1545968319868719. Epub 2019 Aug 22. PMID 31434537